CLINICAL TRIAL: NCT05661942
Title: Diltiazem in the Treatment of Atrial Fibrillation or Atrial Flutter With Rapid Ventricular Rate (AFF RVR): Comparing Calcium Pre-treatment vs Placebo in Prevention of Diltiazem Induced Hypotension
Brief Title: Diltiazem in the Treatment of Atrial Fibrillation or Atrial Flutter With Rapid Ventricular Rate
Acronym: AFFRVR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00107053; 22.135 (Other: Advocate Aurora Health Care)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation With Rapid Ventricular Response; Hypotension Drug-Induced
Keywords: diltiazem; calcium
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcium pre-treatment (Active Comparator): Calcium gluconate 1 gram/100ml 0.9% NaCl or 100ml 0.9% NaCl
  Interventions: Drug: Calcium pre-treatment
- Placebo (Placebo Comparator): diluent (NS) vials
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcium pre-treatment — The intervention is Calcium gluconate 1 gram/100ml 0.9% NaCl or 100ml 0.9% NaCl) over 5 minutes.
  Arms: Calcium pre-treatment
Other: Placebo — Placebo/ no calcium pre-treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see how well calcium pre-treatment works for decreasing incidence of drug-induced hypotension after diltiazem administration for treatment of atrial flutter with rapid ventricular rate.

DETAILED DESCRIPTION:
Non-dihydropyridine calcium channel blockers(CCB) are routinely used in the treatment of atrial fibrillation or flutter with rapid ventricular response (AFF with RVR); however, their use can be limited by drug-induced hypotension. This drug induced hypotension limits and complicates CCB use in the treatment of AFF with RVR. Calcium pre-treatment with calcium channel blocker administration has been studied extensively with verapamil administration in preventing drug induced hypotension however, similar studies evaluating calcium pretreatment with diltiazem administration in the prevention of drug-induced hypotension are limited.

The purpose of this study is to compare the relative efficacy and safety for calcium pretreatment with diltiazem in the treatment of AFF with RVR in preventing drug-induced hypotension. This prospective, randomized double-blinded study will evaluate patients who present to the emergency department at Advocate Christ Medical Center with a diagnosis of AFF with RVR with ventricular rate greater than or equal to 120 beats per minute from IRB approval to June 1, 2024. Via simple randomization, patients will be administered calcium pretreatment versus control prior to diltiazem administration. Calcium gluconate 1 gm or 100 mL of normal saline will be administered as an intravenous infusion over 5 minutes followed by bolus diltiazem 0.25 mg/kg IV push (with a 20 mg max) with repeat diltiazem bolus dose after 15 minutes if rate control not achieved 0.35mg/kg IV push. Calcium gluconate will not be administered with repeat doses of diltiazem. Weight-based dosing of diltiazem was most utilized, though some providers may elect to modify based on the clinical scenario. The primary outcome will be the mean difference in systolic blood pressure evaluated at 5 and 15 minutes after administration of diltiazem bolus. Secondary outcomes include decrease in heart rate, conversion to sinus rhythm, and adverse effects of medication administered.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years or older
* Able to provide informed consent
* Primary diagnosis AFF with RVR greater than or equal to 120 bpm

Exclusion Criteria:

* Pregnancy defined as a positive urine HCG
* Hemodynamically unstable patients (SBP <90, MAP <65)
* Stated history of systolic heart failure with reduced ejection fraction (<40%) or evidence of acute heart failure or reduced EF (peripheral edema, JVD, pulmonary edema) on clinical exam or bedside echo
* Patients with left ventricular assist device
* Sinus node dysfunction or preexcitation with accessory pathway (known diagnosis of SVT, WPW or sick sinus syndrome. Delta waves or other evidence of accessory pathway on EKG)
* 2nd or 3rd degree atrioventricular block
* Allergy or sensitivity to any study drugs
* Previously enrolled in this trial during a different patient encounter
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Cirone, MD, Principal Investigator — Advocate Aurora Health (AAH)
Locations (1):
- Advocate Christ Medical Center Emergency Department (ACMC ED), Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium Pre-treatment | Placebo
Started | 46 | 46
Completed | 44 | 39
Not Completed | 2 | 7
Not completed — Nine patients were excluded due to change in hemodynamic status and consent withdrawal. | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Pre-treatment | Placebo | Total
Number analyzed (Participants) | 44 | 39 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9545 (10.9395) | 68.6923 (11.3721) | 67.7711 (11.1107)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 24 | 16 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 39 | 83
Weight (kg) [Median (Inter-Quartile Range); unit: kilograms] | 87.1000 [73.4000 to 114.4000] | 90.1500 [79.2000 to 111.1500] | 87.3000 [75.4000 to 114.3000]
Height (cm) [Median (Inter-Quartile Range); unit: centimeters] | 167.6000 [160.0000 to 177.8000] | 172.7000 [165.1000 to 181.6000] | 170.2000 [162.6000 to 180.3000]
On rate Control Medicine (yes/no)? [Count of Participants; unit: Participants]
  Yes | 13 | 16 | 29
  No | 31 | 23 | 54
Which Rate Control Agent? [Count of Participants; unit: Participants]
  Metroprolol | 0 | 2 | 2
  Diltiazem | 10 | 10 | 20
  Digoxin | 1 | 2 | 3
  Other | 2 | 2 | 4
  Not on Rate Controlled Agent | 31 | 23 | 54
On Rhythm Medication for PTA? [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 44 | 38 | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Systolic Blood Pressure
Description: Mean difference in systolic blood pressure after administration of diltiazem bolus. Monitors were set to obtain an automated full set of vitals every 5 minutes after administration of diltiazem.
Time Frame: Baseline to 5 Minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
mmHg | -11.7500 (15.7689) | -19.5385 (16.1259)

2. Primary Outcome: Mean Difference in Systolic Blood Pressure
Description: Mean difference in systolic blood pressure evaluated after administration of diltiazem bolus. Monitors were set to obtain an automated full set of vitals every 5 minutes after administration of diltiazem.
Time Frame: Baseline to 10 Minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
mmHg | -7.8182 (14.4484) | -16.2564 (15.0660)

3. Primary Outcome: Mean Difference in Systolic Blood Pressure
Description: as for outcome 1
Time Frame: Baseline to 15 Minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
mmHg | -7.2273 (14.1994) | -13.6667 (16.1267)

4. Secondary Outcome: Mean Change in Heart Rate
Description: Mean difference in heart rate evaluated after administration of diltiazem bolus. Monitors were set to obtain an automated full set of vitals every 5 minutes after administration of diltiazem.
Time Frame: Baseline to 5 Minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
beats per minute | -37.8864 (21.5355) | -36.2564 (20.6687)

5. Secondary Outcome: Mean Change in Heart Rate
Description: as for outcome 4
Time Frame: Baseline to 10 Minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
beats per minute | -43.9545 (19.6551) | -35.0000 (21.5174)

6. Secondary Outcome: Mean Change in Heart Rate
Description: as for outcome 4
Time Frame: Baseline to 15 Minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
beats per minute | -43.1136 (19.1860) | -33.7949 (22.2405)

7. Secondary Outcome: Heart Rhythm at 5 Minutes
Description: Heart rhythm category after 5 minutes of initial diltiazem administration for treatment of AFF with RVR.
Time Frame: Baseline to 5 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
Participants
  AFF | 36 | 29
  AFF RVR | 7 | 9
  NSR | 1 | 1

8. Secondary Outcome: Heart Rhythm at 15 Minutes
Description: Heart rhythm category after 15 minutes of initial diltiazem administration for treatment of AFF with RVR.
Time Frame: Baseline to 15 Minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Calcium Pre-treatment | Placebo
Number analyzed (Participants) | 44 | 39
Participants
  AFF | 36 | 27
  AFF RVR | 6 | 10
  NSR | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the 5 minutes, 10 minutes, and 15 minutes intervals after initiation of diltiazem infusion by the emergency department pharmacy staff associated with this study.
Arm/Group | Calcium Pre-treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/39
Other Adverse Events (participants affected / at risk) | 5/44 | 2/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Pre-treatment (N=44) | Placebo (N=39)
hypotension (General disorders) | 1 (1) | 1 (1)
extravasation via Calcium Gluconate (General disorders) | 1 (1) | 0 (0)
ringing in ears/chest pressure (General disorders) | 2 (2) | 1 (1)
extravasation via CCB (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations: this was a single-center study with a relatively small sample size, which may limit generalizability. There was variability in diltiazem dosing amongst providers. Additionally, variability in provider practice and in dosing and timing of administration was present with the use of magnesium sulfate for atrial flutter with rapid ventricular rate. The timing and dose of magnesium administration was not protocolized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT05661942/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT05661942/ICF_000.pdf